CLINICAL TRIAL: NCT00056082
Title: A Study to Identify Biomarker Modulation by a Cyclooxygenase-2 (COX-2) Inhibitor in Breast Tissue of Premenopausal Women at High Risk for Estrogen Receptor Negative (ERN) Breast Cancer
Brief Title: Celecoxib in Preventing Breast Cancer in At-Risk Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carol Fabian, MD, Director, Breast Cancer Prevention Unit, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KUMC-HSC-8919-02; CDR0000271935 (Registry Identifier: PDQ (Physician Data Query)); N01-CN-15135 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celecoxib 400 mg bid (Experimental): Celecoxib 400 mg bid
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — Celecoxib daily for 12 months
  Other Names: Celebrex

SUMMARY:
RATIONALE: Chemoprevention therapy uses certain drugs to try to prevent the development or recurrence of cancer. Celecoxib may be effective in preventing breast cancer in at-risk women.

PURPOSE: Phase II trial to study the effectiveness of celecoxib in preventing breast cancer in premenopausal women who are at risk of developing cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the change in proliferation in benign breast epithelial cells as measured by Ki-67/MIB-1 in premenopausal women at high risk for estrogen receptor-negative breast cancer treated with celecoxib.
* Determine the feasibility of this regimen by dropout rate of these patients during 12 months of treatment and compliance.
* Determine the proportion of these women likely to express cyclooxygenase-2 protein (COX-2) in at least 10% of benign ductal epithelial cells.
* Compare the success rate of obtaining adequate ductal epithelial cells by random periareolar fine needle aspiration (FNA) and ductal lavage in these patients before vs after 12 months of a prevention intervention.
* Assess pain associated with FNA and ductal lavage in these women.
* Correlate, if possible, serum proteomics pattern with cytologic assessment and mammographic density at baseline and at 12 months in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral celecoxib twice daily. Treatment continues for 12 months in the absence of clinical evidence of cancer confirmed by biopsy or unacceptable toxicity.

Patients are assessed at baseline and at 12 months for mammographic breast density, serum hormone levels, and serum IGF-1/IGFBP-3. Patients undergo ductal lavage or fine needle aspiration for assessment of supernatant proteomics and breast biomarkers.

Patients are followed at 2 weeks and then annually for 5 years.

PROJECTED ACCRUAL: A total of 110 patients will be accrued for this study within 10-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Increased risk for breast cancer on the basis of at least 1 of the following criteria:

  * Five-year Gail risk at least 1.7% or a calculated risk at least 5 times the average for age group

    * 20-29 years old - calculated 5-year Gail risk is at least 0.1%
    * 30-39 years old - calculated 5-year Gail risk is at least 1.0%
    * 40 and over - calculated 5-year Gail risk is at least 1.7%
  * Known BRCA1/BRCA2 mutation carrier
  * Family history consistent with hereditary breast cancer, as defined by any of the following circumstances:

    * At least 4 relatives with breast cancer at any age
    * At least 2 first-degree relatives diagnosed with breast cancer at age 50 or younger
    * Breast and ovarian cancer diagnosed in the same relative
    * At least 2 occurrences of breast cancer and 1 occurrence of ovarian cancer at any age in the same family
  * Prior biopsy exhibiting atypical hyperplasia, lobular cancer in situ, ductal carcinoma in situ (DCIS)*, or invasive cancer** NOTE: *If DCIS or T1a or T1b disease was found, at least 2 months must have elapsed since prior surgery and/or radiotherapy to the involved breast

NOTE: **Prior invasive cancer (T1c, T2, or T3) must have been diagnosed at least 2 years before study and be estrogen receptor-negative, node negative

* Must have had a random periareolar fine needle aspiration successfully performed within the past 3 months, with at least 1,000 cells on cytology slide and 3 additional slides for biomarker analysis (1 with at least 500 cells for Ki-67 and 2 with at least 100 ductal cells for estrogen receptors and COX-2)
* Hormone receptor status:

  * Estrogen receptor negative

PATIENT CHARACTERISTICS:

Age

* 18 to 55

Sex

* Female

Menopausal status

* Premenopausal, defined as menstrual periods estimated to occur every 21 to 35 days over the past 6 months

Performance status

* Not specified

Life expectancy

* At least 5 years

Hematopoietic

* Absolute granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* No bleeding diathesis within the past year

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* Albumin at least 3.0 g/dL
* AST and ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* No severe liver disease requiring treatment

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No high blood pressure not controlled by medication
* No history of angina
* No history of cardiovascular disease
* No history of deep vein thrombosis

Pulmonary

* No history of pulmonary embolism

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergy to sulfa, COX-2 inhibitors, or nonsteroidal anti-inflammatory drugs (NSAIDs)
* No history of an ulcer requiring treatment
* No history of ulcerative colitis
* No inflammatory bowel disease
* No body mass index > 33
* No history of diabetes
* No prior metastatic malignancy of any kind
* No complications of alcoholism requiring hospitalization
* No concurrent asthma being treated

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 6 months since prior chemotherapy

Endocrine therapy

* At least 6 months since prior antihormone therapy (e.g., selective estrogen-receptor modulators or aromatase inhibitors)
* Anticipated use of oral or IV corticosteroids must be less than 2 weeks per year
* No change (stop or start) in hormonal therapy within the past 6 months (e.g., estrogen, progesterone, oral contraceptives, or fertility agents)

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the contralateral breast involved in the study treatment

Surgery

* See Disease Characteristics

Other

* At least 3 weeks since prior aspirin, rofecoxib, celecoxib, other COX-2 inhibitors, or NSAIDs
* No concurrent anticoagulants
* No other concurrent NSAIDs
* No chronic angiotensin-converting enzyme inhibitors
* No chronic furosemide*
* No chronic fluconazole*
* No chronic lithium NOTE: *Occasional concurrent use allowed

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2003-01; Primary Completion 2008-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J. Fabian, MD, Study Chair — University of Kansas
Locations (3):
- United States (3):
  - Lynn Sage Comprehensive Breast Center at Northwestern Memorial Hospital, Chicago, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No
Global results will be published